CLINICAL TRIAL: NCT01155089
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Anastrozole 1 mg Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Anastrozole 1 mg Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANAS-T1-PVFD-1
Record Dates: First submitted 2010-06-28; First posted 2010-07-01 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anastrozole — 1 mg tablet
  Other Names: ARIMIDEX

SUMMARY:
The objective of this study was to prove the bioequivalence of Anastrozole Tablet under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to anastrozole or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-05; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Morrison, D.O., Principal Investigator — Bio-Kinetic Clincial Applications
Locations (1):
- Bio-Kinetic Clinical Applications, Springfield, Missouri, United States